CLINICAL TRIAL: NCT06610058
Title: Effects of Instrument Assisted Soft Tissue Mobilization on Healthy Tissue Regarding Range of Motion and Lower Extremity Power
Brief Title: Effects of Instrument Assisted Soft Tissue Mobilization Regarding Range of Motion and Lower Extremity Power
Acronym: (IASTM)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Marschner (Other)
Collaborators: Minot State University (Other)
Responsible Party: Sponsor-Investigator, Beth Marschner, Assistant Professor, Minot State University
Organization: Minot State University (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 2428
Record Dates: First submitted 2024-09-18; First posted 2024-09-24 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-09

CONDITIONS: Healthy
Keywords: Instrument Assisted Soft Tissue Mobilization; Range of Motion; Lower Extremity Power; Vertical Jump; Horizontal Jump

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- IASTM First (Experimental): This arm of the study received IASTM treatment on the first day and the wait/control on the second day of the study
  Interventions: Other: Instrument Assisted Soft Tissue Mobilization first Control second
- Wait/control First (Experimental): This arm of the study waited (was the control) on the first day and received IASTM treatment on the second day of the study.
  Interventions: Other: Control first Instrument Assisted Soft Tissue Mobilization second

INTERVENTIONS:
Other: Instrument Assisted Soft Tissue Mobilization first Control second — Instrument assisted soft tissue mobilization was utilized first on day one and wait-control was completed on second day.
  Arms: IASTM First
Other: Control first Instrument Assisted Soft Tissue Mobilization second — This intervention involved waiting for 20 minutes between pre-test and post-test on day one and having Instrument Assisted Soft Tissue Mobilization on day two.
  Arms: Wait/control First

SUMMARY:
The goal of this clinical trial is to study the effects of instrument assisted soft tissue mobilization (IASTM) in healthy adult volunteers. The main questions it aims to answer are:

* Does IASTM treatment have an effect on range of motion (ROM) as measured in the hip, knee and ankle?
* Does IASTM treatment have an effect on lower extremity power? Researchers will compare pre-test and post-test IASTM treatment intervention data to the pre-test and post-test data of the no treatment control intervention to see if IASTM works to change range of motion and/or lower extremity power.

Participants will:

* Complete a questionnaire on medical history and injury background
* Have hip, knee and ankle range of motion (ROM) measurements taken on both lower extremities using a goniometer
* Complete three trials of vertical jump testing using a Fleage Floor standing vertical jump measurement tester with one warm up first
* Complete three trials of horizontal jump testing using a Woanger 12'x2.5' long jump mat and verified by a secondary measure using a tape measure with one warm up first
* Be randomly assigned to either IASTM first treatment group or the wait/control first group
* Receive IASTM treatment techniques including application of emollient to the skin to reduce friction on the surface followed by scanning the hamstrings, quadriceps, gastroc/soleus complex, and Achilles tendon using the HG8-Scanner tool for 15 strokes in each direction. Then the concave tool corresponding to the size of the structure being treated will be used (HG6-Large Multi-Curve, HG5-Medium Multi-Curve, HG4-Small Multi-Curve) for 15 strokes in each direction.
* Simply wait for 20 minutes (the duration of time treatment with IASTM would require) when completing the control treatment.
* Complete hip, knee and ankle range of motion and vertical and horizontal jump measure testing at the end of the first session.
* Return within fourteen days after the first session in order to undergo the opposite experience (IASTM first means wait/control second and vice versa).
* Undergo the same baseline pre-test measurements for range of motion and vertical and horizontal jump measure testing as the first session.
* Experience the opposite treatment for the same time period as the first session.
* Undergo the post-test range of motion and vertical and horizontal jump measure testing at the end of the second session for data comparison.

DETAILED DESCRIPTION:
No further information to note than what is described in the summary or elsewhere

ELIGIBILITY:
Inclusion Criteria:

* Individuals from a small regional university student body, faculty and staff may choose to volunteer to participate in this study.

Exclusion Criteria:

* Acute spinal cord injury with neurological deficits
* Neurological disorders
* Acute lower extremity injury such as sprain or strain
* Acute lower extremity pain causing gait deviation
* Any type of lower extremity fracture within the past 12 months
* Lumbar disc pathology with radicular symptoms
* Use of blood thinning or clotting medications
* Known connective tissue disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2024-01-08 (Actual); Primary Completion 2024-02-29 (Actual); Study Completion 2024-02-29 (Actual)

PRIMARY OUTCOMES:
Range of Motion | From baseline to end of session at one hour
  Bilateral hip flexion, extension and abduction, knee flexion and extension, ankle plantarflexion, dorsiflexion, inversion and eversion range of motion measurements were taken in supine or prone (whichever was appropriate) using a goniometer.
Lower Extremity Power Horizontal Jump | From baseline to end of session at one hour
  Lower extremity power was measured by completing three trials of horizontal jump testing using a Woanger 12'x2.5' long jump mat with the distance verified by a secondary measure using a tape measure with one warm up first and 90 seconds to recover between each jump.
Lower Extremity Power Vertical Jump | From baseline to end of session at one hour
  Lower extremity power was measured by completing three trials of vertical jump testing using a Fleage Floor standing vertical jump measurement tester with one warm up first and 90 seconds to recover between each jump.

CONTACTS AND LOCATIONS:
Overall Officials: Beth Marschner, DPT, Principal Investigator — Minot State University
Locations (1):
- Minot State University, Minot, North Dakota, United States

IPD SHARING:
Plan to Share IPD: No
The individual participant data is not the main focus of this study. The overall findings of the study with the larger number of participants to look at the trend is what will be shared (presented or published). The IRB proposal for this study included confidentiality of each individual participant as that will be maintained, but the global findings are what will be shared after data analysis for comparison.